CLINICAL TRIAL: NCT03819829
Title: Blood Sampling of Healthy Volunteers for Immunological Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B18HIR
Record Dates: First submitted 2018-12-13; First posted 2019-01-29 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Other): Blood sample
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample

SUMMARY:
This protocol will be used to collect crucial components of the immune system from healthy volunteers for the characterization of immune cells in fresh blood. A pipeline has been set up for comprehensive immune phenotyping of both lymphoid and myeloid cells within 24 hours after blood withdrawal.

DETAILED DESCRIPTION:
In order to properly compare the immunobiology of healthy volunteers to (advanced) cancer patients, the investigators use age-matched controls with no history of cancer and no potentially interfering medication.

Healthy volunteers will be asked to donate 5 tubes of blood

ELIGIBILITY:
Inclusion Criteria:

* Age above 35 years
* Written informed consent
* No history of cancer
* No use of systemic immunosuppressive medication (eg. corticosteroids). Local use of corticosteroids (eg. topical or inhalation) is allowed.

Exclusion Criteria:

* Fever 14 days before blood withdrawal
* Donated blood for the same program within the last 2 years
* Pregnancy

Min Age: 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
The number of immune cells, both lymphoid and myeloid, present in the blood of healthy individuals, assessed by flow cytometry, as well as cytokine expression and transcriptome profiles of these cells | assessed up to 12 months
  the number of lymphoid and myeloid immune cells present in the blood of healthy individuals using flow cytometry, assessing the cytokine expression of these cells in healthy individuals using ELISA cytokine assays, and assessing gene expression of these cells using single cell transcriptomics analyses using droplet-based single cell RNA sequencing.

SECONDARY OUTCOMES:
Immunophenotyping of both myeloid and lymphoid cells in healthy individuals | assessed up to 12 months
  Immunophenotyping of both myeloid and lymphoid cells in healthy controls to gain insights in immunological defects and immune evasion in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: M Kok, MD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be determined